CLINICAL TRIAL: NCT01143779
Title: FLT-PET as an Imaging Biomarker in Patients Receiving the Combination of Cell Cycle Inhibitors Temsirolimus, Topotecan, and Bortezomib
Brief Title: FLT-PET as an Imaging Biomarker With Temsirolimus, Topotecan, and Bortezomib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0658
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2022-01-04 (Actual); Status verified 2022-01

CONDITIONS: Advanced Cancer
Keywords: Advanced Malignancy; FLT-PET Scan; [F-18]-fluoro-L-thymidine; FLT; Positron emission tomography; PET; Imaging Biomarker; Temsirolimus; Topotecan; Bortezomib
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FLT-PET (Experimental): FLT-PET scan uses the FLT solution (dosage of FLT in range between 1 and 10 mCi) with imaging performed 60-90 minutes after FLT intravenous injection.
  Interventions: Drug: FLT-PET

INTERVENTIONS:
Drug: FLT-PET — FLT-PET scan uses the FLT solution (dosage of FLT in range between 1 and 10 mCi) with imaging performed 60-90 minutes after FLT intravenous injection.
  Other Names: [F-18]-fluoro-L-thymidine; positron emission tomography

SUMMARY:
The goal of this clinical research study is to learn if an imaging solution, [F-18]-fluoro-L-thymidine (FLT), when used with a positron emission tomography (PET) scan, can help doctors to better see changes in the growth of tumors in the body. Researchers want to learn if FLT-PET scans can show an early response to chemotherapy.

DETAILED DESCRIPTION:
FLT-PET Scan:

An FLT-PET scan uses the FLT solution, which contains a small amount of radioactive material, to help locate cancer cells inside the body. This scan may help doctors find solid tumors as well as learn if these tumors are growing and how fast they are growing. This information could be used to help predict if the cancer will respond to treatment.

Study Visits:

Within 2 weeks before Day 1 of Cycle 1 and between Days 19 and 21 of Cycle 1, you will have a FLT-PET scan.

For at least 4 hours before the FLT-PET scan, you must not eat or drink anything. You will receive the FLT solution by vein. The FLT solution is a mildly radioactive material. The radioactive nature of the solution allows the scanner to "see" it in certain places in your body. After the injection, you will need to rest quietly until it is time for the scan. The amount of rest time may vary, but be prepared to wait for about 60 minutes. During the scan, you will lie flat on your back on a table. After the solution is injected into a vein, the PET scanner takes pictures of the radioactive solution as it moves through the body and collects at various sites in the body. By watching how the solution travels through the body and studying where the solution collects, researchers can learn the status of disease in the body. The scan itself may last about 40-60 minutes.

Your vital signs (blood pressure, heart rate, temperature, and breathing rate) will be measured before each injection of the FLT solution, 30 minutes after each injection, and before each PET scan. You will be allowed to leave 30 minutes after your scan, if your vital signs are acceptable.

Length of Study:

You will be off this study after the second FLT-PET scan. You will be taken off study early if you have intolerable side effects or the study doctor thinks it is in your best interest.

This is an investigational study. The FLT solution is not FDA approved or commercially available. At this time, FLT solution is only being used in research.

Up to 5 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients enrolled on Protocol 2008-0425: "A Phase I Study of Temsirolimus, Topotecan, and Bortezomib in Patients with Advanced Malignancy" or Protocol 2012-0061: "A Phase I Trial of Bevacizumab, Temsirolimus Alone and in Combination with Valproic Acid or Cetuximab in Patients with Advanced Malignancy" are eligible. These patients must have met the inclusion and exclusion criteria for that protocol.
2. Women of child-bearing potential (as defined as women who are not post-menopausal for 12 months or who have had no previous surgical sterilization) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days after the last dose.
3. Ability to understand and the willingness to sign a written informed consent document.
4. Patients must be at least 18 years of age

Exclusion Criteria:

1. Pregnant or breast-feeding women.
2. History of hypersensitivity to 3'-deoxy-3'-18F-fluorothymidine (18F- FLT) or any component of the formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Patient Standardized Uptake Value (SUV) | Cycle 1, Day 21
  SUV measured on continuous scale at two specified time points (baseline and post-treatment phase, cycle 1, day 19-21).

CONTACTS AND LOCATIONS:
Overall Officials: Sarina Piha-Paul, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org